CLINICAL TRIAL: NCT01830894
Title: Evaluation and Correlation Between the Disruption in Blood-brain-barrier and the Development of Secondary Brain Edema Associated With Brain Damage by Using MRI in Patients With Various Types of Intra-cranial Bleeding
Brief Title: Feasibility Study of New MRI Protocol in Assessing Early Blood Brain Barrier Disruption (BBBD)in Related to Delay Brain Edema
Acronym: BBBD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Sagi Harnof, M.D., Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-12-9889-SH-CTIL
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-03

CONDITIONS: Intra Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- spontaneous ICH bleeding (Experimental): An initial Baseline MRI is to be done within 6-24 hours from the bleeding. second MRI which serves as review - on the 3rd -5th day after bleeding
  Interventions: Device: MRI
- chronic sub dural bleeding (Experimental): An initial Baseline MRI is to be done at the time of diagnosis. second MRI which serves as review -within two weeks.
  Interventions: Device: MRI
- acute sub-dural bleeding (Experimental): An initial Baseline MRI is to be done within 6-24 hours from the bleeding. second MRI which serves as review - within two weeks.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — 3 MRI on different times during the study for each arm.
  Other Names: BBB disruption detection algorithm using Gad enhanced MR

SUMMARY:
MRI research Group in the Advanced Technology Center of the Sheba Medical Center has developed an innovative methodology based on leakage (extravasation) contrast agent that allows to map the entire brain with high resolution and high sensitivity to check and describe disorders BBB (blood brain barrier).

The aim of the current study is to evaluate the feasibility of the BBB disruption detection method to predict delayed peri - hemorrhage edema.

DETAILED DESCRIPTION:
Research's Protocol:

Evaluation and Correlation between the disruption in blood-brain-barrier and the development of secondary brain edema associated with brain damage by using MRI in patients with various types of intra-cranial bleeding .

Research team:

Main (Primary researcher):

Sagi Harnof MD , Neurosurgery department, Sheba medical center, Tel Hashomer

Secondary researchers:

Prof. David Tanne (M.D), Neurology department .

Dr. Yael Mardor (PhD), Advanced technology department.

Dr. Oded Goren (M.D), Neurosurgery department.

Dr. Masswadeh Ahmad (M.D), Neurosurgery Department.

Background :

Spontaneous brain hemorrhage is one of the most difficult issues in strokes concept regarding underlying pathology, reasons and treatment.

Etiology:

* General prevalence of about approximately 10-15% in all strokes.
* Mortality and morbidity associated with it are the most severe with mortality rates of up to 50-60%.

There are various pathologies thought to be responsible for bleeding, most commonly known to be :

hypertension, Angiopathies, amyloidotic or vascular problems and space occupying lesions.

Treatment process that takes place is very limited and most patients are treated only conservatively.

Cytotoxic brain edema that develops around the bleeding results usually from local cell damage and local pressure. It usually increases in the first days after bleeding and is considered to be one of the main causes of deterioration after cerebral hemorrhage .

Sub-dural cerebral hemorrhage is a common disease due to traumatic injury, often with serious consequences.

Regarding the natural history of subdural bleeding, not only It's believed to be difficult predicting the bleeding's course, but the risk to induce cerebral edema and later on to develop into chronic sub Dural bleeding is unpredictable as well .

Nevertheless chronic sub-dural bleeding is one of the most common cases seen in neurosurgery practice, But worthy to notify that only little is known about the pathogenesis of the disease, appearance of symptoms , preferable time for drainage and its complications .

Although hasn't been contributing much in clinical evaluation of stoke, MRI has a growing importance in the field of stroke lately .

In a previous neuro-imaging research that included patients after ischemic stroke it was shown that with an innovative methodology based on leakage extravasation) contrast agent in MRI which allows to map the entire brain with high resolution, we can easily evaluate the sensitivity disorder in BBB .

In 27% of patients who showed no anomalies at BBB in normal MRI, calculated maps with late leakage showed significant volumes of BBB opening ischemic areas.

MRI research Group in the Advanced Technology Center of the Sheba Medical Center has developed an innovative methodology based on leakage (extravasation) contrast agent that allows to map the entire brain with high resolution and high sensitivity to check and describe disorders BBB.

Data Acquisition:

MRI will be performed using the General Electric (GE) T3.0/1.5 with a standard head coil of 8 channels.

MRI scans will include high-resolution spin-echo T1-weighted MRI , acquired before and at several time points after injection (1, 12, 20, 23, 30, 70 minutes after injection).

T1-MRI may be done with Echo Time (TE) / Repetition Time (TR) = 22/240 ms, field of view 26 x 19.5 inch, 5/0.5 mm slice thickness and 512x512 - pixels.

To notify : T1-MRI data is acquired simultaneously with any conventional imaging protocol accepted at Sheba Medical center by routine practice. (Sheba's routine).

Type of study:

A prospective feasibility study performed on a group of patients with cerebral hemorrhage.

The purpose of the study:

1. Assess the ability to characterize quantitatively the BBB disruption around cerebral hemorrhage.
2. Find a correlation between the degree of BBBD immediately after bleeding and cerebral edema 3-5 days after bleeding.
3. Search for clinical correlation between the degree of BBBD immediately after the bleeding and the clinical course that follows it later on.

Methods:

This is a prospective study aimed to test the feasibility of using BBBD protocol in MRI in order to predict the development of edema and clinical deterioration.

Course of the experiment:

Once the -on call- neurosurgery resident is notified about a patient with spontaneous ICH he would contact any of the researchers to begin the screening process for participation in the study. Patients who had undergone intracranial hemorrhage (ICH) that was discovered in the past twelve hours will undergo a screening process performed by any of the researchers in order to determine whether or not they meet the inclusion criteria. Such patients may arrive from the emergency room, intensive care unit or any of the other wards in the hospital.

3. An initial Baseline MRI is to be done:

1. for spontaneous ICH bleeding - within 6-24 hours from the bleeding.
2. for chronic sub dural bleeding - at the time of diagnosis .
3. for acute sub-dural bleeding - within 6-24 hours from the bleeding.

It should be emphasized that the purpose of the MRI is to assess the extent of BBBD and is intended for research purposes only. This MRI protocol does not allow complete diagnostic assessment. .

Whether the patient needs an accompanying doctor while in MRI or not, is solely determined by a researcher, depending on the patient's clinical situation.

4. Clinical follow-up : neurological status, registration of National Institutes of Health Stroke Scale (NIHSS questionnaire).

a- for spontaneous bleeding - Daily monitoring & registering National Institutes of Health Stroke Scale (NIHSS) for five consequent days. Additional clinical follow-up will be performed two weeks later.

b- for chronic or acute sub-dural bleeding follow up visit after 14 days.

5. second MRI which serves as review :

1. for spontaneous intra-cranial bleeding: on the 3rd -5th day after bleeding.
2. For chronic sub Dural bleeding : within two weeks.
3. For acute sub Dural bleeding: within two weeks.

   6. Two months later, third MRI will be reviewed for all types of bleeding.

   7. Result - Analysis of the outcomes as follows:

   Search correlation between BBBD and clinical status. Search BBBD correlation with hematoma growth.

   Search correlation between BBBD and the development of cerebral edema.

   Search correlation between BBBD and growth process of Chronic Subdural Hematoma (CSDH)

   Search correlation between BBBD and the drainage of CSDH.

   Search correlation between BBBD while Acute Subdural Hematoma (ASDH) is converted to CSDH.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years.
* patient is able to sign the informed consent form.
* Spontaneous brain hemorrhage ICH in the last12 hours ( pre- admission,or sub- dural bleeding (whether acute or chronic ).

Exclusion Criteria:

* The patient meets a contraindication to undergo MRI.
* The patient is too unstable to undergo MRI
* The patient is a candidate for surgery within 24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
delayed peri - hemorrhage edema as a relation to early BBB disruption | 1 week
  early BBB disruption will be calculated from Gad enhanced magnetic resonance (MR) and a correlation to late volume of edema as calculated using 3D methods will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Sagi Harnof, MD, Principal Investigator — Neurosurgery department, Sheba medical center, Tel Hashomer
Locations (1):
- Sheba medical center, Tel Hashomer, Ramat Gan, Israel